CLINICAL TRIAL: NCT05818969
Title: Effects of Hypnosis Therapy on Outcomes in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2.0 - 20203698
Record Dates: First submitted 2023-03-15; First posted 2023-04-19 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Opioid Use
Keywords: Hypnosis; Total Knee Arthroplasty; Total Knee
MeSH Terms: conditions — Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Therapy Group (Experimental): Experimental: Hypnosis Therapy Group
  Patients will receive questionnaires to establish their attitudes/beliefs toward hypnosis, baseline pain, anxiety, & knee function. 7 days prior to surgery, they will receive a pre-recorded video (-19 min) of guided hypnosis to be watched at least 1x/day, until surgery. Postoperative course will be otherwise completely standard of care, including a clinic visit at 10 days after surgery, where they will be given these same questionnaires. Patients will answer them again on postoperative day 49, constituting a study endpoint. Access to pain medication & study doctor will be the same as any total knee arthroplasty regardless of study participation.
  Interventions: Behavioral: Hypnosis Therapy
- Control Care Group (No Intervention): No Intervention: Control Care Group
  Patients will receive questionnaires to establish their attitudes/beliefs toward hypnosis, baseline pain, anxiety, & knee function. 7 days prior to surgery, they will receive a pre-recorded video (-19 min) of guided information to be watched at least 1x/day, until surgery. Postoperative course will be otherwise completely standard of care, including a clinic visit at 10 days after surgery, where they will be given these same questionnaires. Patients will answer them again on postoperative day 49, constituting a study endpoint. Access to pain medication & study doctor will be the same as any total knee arthroplasty regardless of study participation.

INTERVENTIONS:
Behavioral: Hypnosis Therapy — Pre-recorded hypnosis therapy audio recording with accompanying visual of a calming ocean scene to be played at least once daily for 7 days preoperatively.
  Other Names: Hypnotherapy
  Arms: Hypnosis Therapy Group

SUMMARY:
The purpose of this study is to collect information to evaluate the role of the psychogenic component of pain induced by anxiety on postoperative outcomes in major orthopaedic surgery and to determine whether hypnosis therapy provided during the perioperative period will lead to decreased use of opioid therapy. Patients are randomly assigned to one of two treatment groups: (I) usual care, or; (II) hypnotherapy treatment. Patients have an equal chance of being assigned to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary knee arthritis, in need of a total knee arthroplasty.
* The ability to read, speak, and understand English
* The ability and willingness to use a web-based application (OBERD) on a smartphone, pad/tablet, or computer
* 18 years of age or older

Exclusion Criteria:

* Revision total knee arthroplasty
* Any knee procedure except a primary knee arthroplasty, since these procedures have shown to result on increased postoperative pain compared to primary surgery
* Patients with active cancer or receiving palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Perioperative Anxiety - Amsterdam Preoperative Anxiety and Information Scale (APAIS) | 7 days prior to surgery, 10 days postoperative day, 49 days postoperative day
  Patient-reported anxiety in the perioperative period

SECONDARY OUTCOMES:
Change in Perioperative Pain - Knee Society Score/ Knee Injury and Osteoarthritis Scores | 7 days prior to surgery, 10 days postoperative day, 49 days postoperative day
  Patient-reported pain in the perioperative period
Change in Opioid Consumption - The Beliefs and Attitudes to Hypnosis Valencia Scale-Client | 7 days prior to surgery, 10 days postoperative day, 49 days postoperative day
  Change in Anxiolytic Consumption
Change in Anxiolytic Consumption - The Beliefs and Attitudes to Hypnosis Valencia Scale-Client | 7 days prior to surgery, 10 days postoperative day, 49 days postoperative day
  Change in Anxiolytic Consumption

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Palumbo, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No